CLINICAL TRIAL: NCT06673836
Title: Comparative Effect of Inclined Treadmill and Dynamic Cycling on Balance and Gait in Children With Hearing Impairment.
Brief Title: Comparative Study of Inclined Treadmill and Dynamic Cycling on Balace in Hearing Impaired Children.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/ASRA GHAFOOR
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Balance Assessment
Keywords: balance; dynamic cycling; gait

STUDY DESIGN:
Intervention Model Description: parallal assignment. it will be randomized controlled study,in which probability convenient sampling will be usd.two groups of hearing impaired children will be randomly divided.
Who Masked: Participant
Masking Description: participant will get separate treatment protocols and possible effort will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic cycling (Experimental): one group will perform dynamic cycling for 6 consecutive weeks,3 days a week for 30 minutes per session.
  Interventions: Device: DYNAMIC CYCLING
- inclined treadmill (Experimental): one group will perform treadmil for 3 days a week with 10 degree inclination for 6 six consecutive weeks.
  Interventions: Device: INCLINED TREAD MILL

INTERVENTIONS:
Device: DYNAMIC CYCLING — Balance Training: Exercises focused on improving coordination and balance, such as standing on one leg, walking on uneven surfaces, or using balance boards.
  Core Strengthening: Strengthening core muscles helps children maintain stability during dynamic movements, such as walking or running.
  Proprioceptive Training: Exercises that improve awareness of the body's position in space, such as obstacle courses or activities that challenge movement coordination.
  Other Names: Balance Training: Exercises focused on improving coordination and balance, such as standing on one leg, walking on uneven surfaces, or using balance boards. Core Strengthening: Strengthening core musc; inclined treadmill training is a powerful tool for addressing the balance and gait challenges faced by hearing-impaired children. Through gradual and progressive training, this intervention helps to s
  Arms: dynamic cycling
Device: INCLINED TREAD MILL — Dynamic Cycling: Refers to the fluctuating nature of movement patterns, often used in therapies like stationary biking or recumbe.nt cycling, where the intensity and resistance vary. Dynamic cycling can also refer to training that involves alternating between high and low-intensity phases or cycling between different positions (sitting, standing) or speeds during the activity
  Other Names: dynamic cyling
  Arms: inclined treadmill

SUMMARY:
Hearing loss is generally identified initially in life leading to difficulties in communication. In children, vestibular dysfunctions can cause a deficit in gross motor development and balance stability. At an early age, delayed gross motor development can cause impairment in the bilateral vestibular system and sensorineural hearing. The children with balance impairment cannot usually participate in physical activities. Running, cycling, hoping and leading to social isolation3. In Pakistan, 2.49% of the population suffers from some disability; the hearing loss population is 7.4%. In Pakistan, hearing loss is more reported in males as compared to females. According to the non-official data, nearly 1.2 in every 1000 Pakistani children suffer from moderate to severe bilateral hearing loss5. In this, 15% population is suffering from profound and nearly 85% from moderate to severe hearing loss.Children who have vestibular dysfunctions may experience many disorders of the vestibular system.Acute unilateral vestibular loss (AUVL) is the most frequent vestibular dysfunction. The etiology of acute unilateral vestibular loss is unknown, but the studies say it may be due to genetic and acquired causes (inflammatory and viral infections). The symptoms include static

DETAILED DESCRIPTION:
This study seeks to provide a detailed understanding of the effects of dynamic cycling and inclined treadmill training on the motor skills of children with hearing impairments through an extensive review of relevant literature, careful data collection, and robust statistical analysis. The findings may assist parents, educators, and healthcare professionals in making informed choices about the most effective therapies to enhance mobility and overall development in children with hearing impairments. Ultimately, this research contributes to pediatric rehabilitation and promotes a holistic approach to addressing the specific needs of children with hearing loss.

ELIGIBILITY:
Inclusion Criteria: children of age 8 to 10 years consistency in hearing impairment ability to understand the command

Exclusion Criteria:

children with any acute or chronic disease recurrent falls history of any MSK disease

-

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic gate index | 10-15 min
  The Dynamic Gait Index was developed by Anne Shumway-Cook (1995) and has been used with older adults to determine their likelihood of falling. Scores of 19 and less are related to falls in older adults. It tests 8 facets of gait and can be used with an assistive device.
CTSIB TEST | 10 min
  The test is the therapist's version of the Computerized Dynamic Post urography which attempts to measure the way that vision, Vestibular and somatosensory interaction allows us to maintain our balance against the forces of gravity. The test was developed by Shumway Cook and Horak in 1986 and further discussed as a clinical tool in 1987 Patients with uncompensated unilateral vestibular deficits have been shown to have difficulty when visual and support surface information are manipulated.

CONTACTS AND LOCATIONS:
Overall Officials: Asra Ghafoor, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strader DB, Wright T, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C. Hepatology. 2004 Apr;39(4):1147-71. doi: 10.1002/hep.20119. No abstract available. PMID 15057920